CLINICAL TRIAL: NCT03300713
Title: MOther-Child Interaction Assessment TRAINING for Pediatricians
Acronym: MOCITRAINING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015_04; 2016-A00540-51 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Child Behavior Disorders; Mother-child Relations; Depression, Postpartum
Keywords: Mass screening; Pediatrician training
MeSH Terms: conditions — Child Behavior Disorders; Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F+ group (Mocitraining program) (Experimental): including 8 pediatricians' clusters. F+ pediatricians will attend a specific training focused on mother-child interactions, maternal psychiatric disorders, particularly PND screening and early interventions for non-psychiatric physician.
  Interventions: Other: MOCITRAINING program
- F- group (usual follow-up) (Sham Comparator): grouping 8 pediatricians' clusters. They will not receive the initial training on early interactional disorders and PND screening
  Interventions: Other: usual follow-up

INTERVENTIONS:
Other: MOCITRAINING program — The program is clinical and psychometric tools for screening for interactions and postpartum psychiatric disorders. The program will expose the existing care arrangements and the different possible orientations of the families according to the identified problem.
  Arms: F+ group (Mocitraining program)
Other: usual follow-up — usual follow-up
  Arms: F- group (usual follow-up)

SUMMARY:
The originality of the MOCITRAINING study lies in the integration of infant and maternal care during the pediatric consultation and the assessment of the impact of this type of care in the short and medium term on The MOCITRAINING program could contribute to improving the quality of parent-child interactions.

ELIGIBILITY:
Inclusion Criteria:

* Each child will be included WITH his biological mother at the first-month visit after birth.
* Age: 1 month + / - 15 days (child), accompanied by his biological mother
* Mother able to read French;
* Signed consent letter after complete information of parents about the MOCITRAINING study, its principle, advantages and disadvantages.

Exclusion Criteria:

* Preterm babies.
* Children from a twin or multiple pregnancy.
* Children with somatic diagnosis explaining the presence of digestive, sleeping or interactional disorders.
* Refusal to participate after clear information about the study;
* Refusal to sign the consent letter;
* Refusal to be informed of a diagnostic hypothesis;
* Participants not covered by the Social Security system;
* Participants incapable of consenting or under legal protection (guardianship or curatorship).

Ages: 23 Days to 37 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3504 (Estimated)
Dates: Start 2017-12-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of pathological Alarm Distress BaBy (ADBB) scores | in 12-month-aged children.

SECONDARY OUTCOMES:
Frequency of pathological Alarm Distress BaBy (ADBB) scores | in 4, 9 and 24 month-aged children
Frequency of digestive disorders | in 4, 9, 12 and 24 month-aged children
  presence/absence of infantile regurgitations and colics
Number of daytime sleep hours | in 4, 9, 12 and 24 month-aged children
Number of nighttime awakenings | in 4, 9, 12 and 24 month-aged children
Scores on maternal self-evaluation scales (Likert scales) | at 12 and 24 months postpartum
  Scores on maternal self-evaluation scales (Likert scales) about parent-child relations (Items concerning comfort and pleasure during interactions)
Frequency of dyads referred for psychiatric or perinatal psychiatric consultations | in 4, 9, 12 and 24 month-aged children
Frequency of maternal psychotropic medication | in 4, 9, 12 and 24 month-aged children

CONTACTS AND LOCATIONS:
Overall Officials: Renaud Jardri, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU, Lille, France

IPD SHARING:
Plan to Share IPD: No